CLINICAL TRIAL: NCT03092544
Title: Investigating Indirect Mechanism of Neuroprotection of Tecfidera® (Dimethyl Fumarate) in RRMS and Progressive Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Multiple Sclerosis Center of Northeastern New York (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BG12-002
Record Dates: First submitted 2016-06-23; First posted 2017-03-28 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- RRMS on therapy (Active Comparator): 18 subjects with a diagnosis of Relapsing Remitting (RRMS) ages 18-55, that are scheduled to begin on dimethyl fumarate
  Interventions: Drug: dimethyl fumarate
- SPMS on therapy (Active Comparator): 18 subjects with a diagnosis of Secondary Progressive (SPMS) ages 25-65 without clinical or MRI evidence of relapse in two years that are scheduled to begin on dimethyl fumarate
  Interventions: Drug: dimethyl fumarate
- SPMS not on therapy (No Intervention): 18 subjects with a diagnosis of SPMS ages 25-65 without clinical or MRI evidence of relapse in two years, that are NOT scheduled to begin on dimethyl fumarate
- Normal Control 1 (No Intervention): 10 normal controls (younger cohort, mean age 38)
- Normal Control 2 (No Intervention): 10 normal controls (younger cohort, mean age 58)

INTERVENTIONS:
Drug: dimethyl fumarate — Active drug
  Other Names: Tecfidera,
  Arms: RRMS on therapy; SPMS on therapy

SUMMARY:
The purposes of this study is to identify types of bacteria that reside in the intestine of healthy individuals and compare them to individuals with Multiple Sclerosis (MS). There has been a lot of research in other autoimmune diseases which has demonstrated the importance of stomach "gut" bacteria because it has an important relationship with the immune system, but this has never been studied in MS patients. In this study investigators aim to show differences in the gut bacteria between healthy individuals and those with MS, to provide a basis for future research studying how diet can affect MS through its effects on the "gut" bacteria.

Additionally, this study will be looking at the effects of dimethyl fumarate on cerebrospinal fluid, plasma and MRI in MS patients taking dimethyl fumarate as compared to those with MS not on dimethyl fumarate or other disease modifying therapy and those who do not have MS (normal controls).

ELIGIBILITY:
Inclusion Criteria:

Inclusion (MS Population Only)

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Male or female subject, age 18-65 (inclusive) at the time of informed consent, with a confirmed diagnosis of multiple sclerosis and meeting multiple sclerosis patient population as specified in section 4/ study design/multiple sclerosis population of this protocol.
2. Subject has the ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
3. Expanded Disability Status Scale (EDSS) score between 0 and 7, inclusive, at screen.

Exclusion (MS Population Only)

General and Medical History Exclusions

1. A MS relapse, as determined by the investigator, that occurred within 90 days prior to screen or the subject has not stabilized from a previous relapse prior to screen visit.
2. Current smoker
3. Any contraindication to having a brain MRI (e.g. pacemaker, MRI-incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed) or contraindication for administration of gadolinium-contrast agents.
4. Clinically significant brain MRI findings other than those related to MS, as judged by the investigator, at screen.
5. Any contraindications to having a Lumbar puncture (LP) (i.e. Aspirin (ASA) greater than 325mg/day, Coumadin, Plavix, decreased platelet count) as determined by the investigator.
6. History of Chronic Urinary Tract Infections, Irritable Bowel Syndrome, Inflammatory Bowel Disease, Diabetes Mellitus or vascular disease as determined by history and investigator decision
7. Evidence or history of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, ulcerative colitis, diabetes mellitus or others) with the exception of MS.
8. History of or current clinically relevant gastrointestinal bleeding or other gastrointestinal diseases or processes that may interfere with the analysis of stool samples per protocol.
9. Any sign of chronic active infection (e.g. urinary tract infection (UTI), bronchitis, hepatitis and tuberculosis) except for those requiring topical medication for treatment (e.g., athletes foot), or screening laboratory evidence consistent with a significant chronic active acute infection requiring systemic treatment. This must be resolved before treatment may commence, (e.g., acute respiratory tract, urinary tract, or gastrointestinal tract infections).
10. Pregnant females; breastfeeding females and/or males of childbearing potential; females of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 28 days after the last dose of dimethyl fumarate use in this protocol. For females of childbearing potential in the dimethy fumarate population; a positive pregnancy test at anytime within the protocol.
11. Known Positive HIV antibody, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody tests indicative of present or prior infection.
12. Any abnormal hematology values or clinical chemistry values judged by the Investigator or Sponsor as clinically significant.
13. Positive purified protein derivative (PPD) skin test or positive quantiferon (QTFN) at screen visit or know history of active tuberculosis not adequately treated.
14. Any malignancy within 5 years, except for basal or Squamous cell skin lesions which have been surgically excised, with no evidence of metastasis.
15. Any clinical, CSF or MRI evidence for Progressive multifocal leukoencephalopathy (PML), from historical MRI or results of the screen MRI.
16. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
17. Subjects participating in or expecting to participate in other interventional clinical trials.
18. Inability or unwillingness to record online dietary questionnaire information as required by protocol
19. History of drug or alcohol abuse (as defined by the investigator) within 2 years prior to screen.

    Exclusion Criteria related to Medication
20. Previous Exposure to dimethy fumarate for disease management at any time in the past.
21. Treatment with methylprednisolone or other systemic corticosteroid for multiple sclerosis relapse or otherwise within 30 days prior to day one of IP administration.
22. Treatment with multiple sclerosis disease modifying therapies as follows:

    * Beta interferons (interferon beta-1a [Avonex® or Rebif®] or interferon beta-1b [Betaseron®], or glatiramer [Copaxone®] within 6 weeks prior to Baseline.
    * Fingolimod (Gilenya®), Teriflunomide (Aubagio®) or washout with accelerated elimination and verification of zero serum levels of teriflunomide prior to day one baseline)
    * Tysabri® (Natalizumab)

      * within 6 months prior to screen OR
      * one month prior to screen if subject has a positive Nabs to Tysabri®
    * Treatment within the past 5 years or current treatment with any of the following agents: cyclosporine, cladribine, that are immunosuppressive (e.g. rituximab, etanercept, cellcept, others), murine protein, T-cell vaccination, plasmapheresis, IV immunoglobulin (IgG) or stem cell transplantation prior to screen.
23. Receipt of any non-live vaccine within the previous 14 days or live vaccine within 30 days prior to first dose of investigational product (IP).
24. Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study medication, whichever is longer.
25. Use of antibiotics for any reason within 3 months of screen.

Inclusion (Normal Control Volunteer Only)

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Normal control volunteer meeting age and co-inhabitant criteria as specified in section 4/ study design/normal control population of this protocol.
2. Subject has the ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.

   Exclusion (Normal Control Population Only)

   General and Medical History Exclusions
3. Current Smoker
4. Any contraindications to having a lumbar puncture (LP) (i.e. ASA greater than 325mg/day, Coumadin, Plavix, decreased platelet count) as determined by the investigator.
5. History of Chronic Urinary Tract Infections, Irritable Bowel Syndrome, Inflammatory Bowel Disease, Diabetes Mellitus or vascular disease as determined by history and investigator decision.
6. Evidence or history of autoimmune disease (e.g., rheumatoid arthritis, systemic lupus erythematosus, ulcerative colitis, diabetes mellitus or others) including the diagnosis of MS or MS symptomatology.
7. History of or current clinically relevant gastrointestinal bleeding or other gastrointestinal diseases or processes that may interfere with the analysis of stool samples per protocol.
8. Any malignancy within 5 years, except for basal or squamous cell skin lesions which have been surgically excised, with no evidence of metastasis.
9. Any sign of chronic active infection (e.g. UTI, bronchitis, hepatitis and tuberculosis) except for those requiring topical medication for treatment (e.g., athletes foot), or screening laboratory evidence consistent with a significant chronic active acute infection requiring systemic treatment. This must be resolved before treatment may commence, (e.g., acute respiratory tract, urinary tract, or gastrointestinal tract infections).
10. Pregnant or breastfeeding females
11. Known Positive HIV antibody, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody tests indicative of present or prior infection.
12. Any abnormal hematology values or clinical chemistry values judged by the Investigator or Sponsor as clinically significant at baseline visit.
13. Other severe acute or chronic medical or psychiatric condition or laboratory abnormalities that may increase the risk associated with study participation or investigational product administration or that may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
14. Inability or unwillingness to record online dietary questionnaire information as required by protocol.
15. History of drug or alcohol abuse (as defined by the investigator) within 2 years prior to baseline.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma samples collected from stable RRMS patients on dimethyl fumarate for their ability to induce changes in neuronal bioenergetics | change from baseline at 6 months treatment with dimethyl fumarate
Change in cerebrospinal (CSF) samples collected from stable RRMS patients on dimethyl fumarate for their ability to induce changes in neuronal bioenergetics | change from baseline at 6 months treatment with dimethyl fumarate
change in levels of neurofilament( NFL) in RRMS patients | at baseline and after 6 months of therapy
change in levels of ceramide sphyngosine and other lipid species in samples collected from patients before and after therapy in CSF samples in RRMS patients | at baseline and 6 months of therapy
changes in microbiota composition consequent to dimethyl fumarate treatment. | 6 months of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Edwards, M.D., Principal Investigator — MS Center of Northeastern NY
Locations (1):
- Multiple Sclerosis Center of Northeastern New York, Latham, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JY, Shen S, Dietz K, He Y, Howell O, Reynolds R, Casaccia P. HDAC1 nuclear export induced by pathological conditions is essential for the onset of axonal damage. Nat Neurosci. 2010 Feb;13(2):180-9. doi: 10.1038/nn.2471. Epub 2009 Dec 27. PMID 20037577
- [Background] Vidaurre OG, Haines JD, Katz Sand I, Adula KP, Huynh JL, McGraw CA, Zhang F, Varghese M, Sotirchos E, Bhargava P, Bandaru VV, Pasinetti G, Zhang W, Inglese M, Calabresi PA, Wu G, Miller AE, Haughey NJ, Lublin FD, Casaccia P. Cerebrospinal fluid ceramides from patients with multiple sclerosis impair neuronal bioenergetics. Brain. 2014 Aug;137(Pt 8):2271-86. doi: 10.1093/brain/awu139. Epub 2014 Jun 3. PMID 24893707